CLINICAL TRIAL: NCT01792258
Title: Procedures, Complications and Follow-up of Percutaneous Tracheostomies in Intensive Care Unit
Brief Title: Procedures and Follow-up of Percutaneous Tracheostomy in Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Professor, University of Genova
Other Study IDs: 53/12
Record Dates: First submitted 2013-02-06; First posted 2013-02-15 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Acute Respiratory Failure; Neurological Disease; Heart Failure
Keywords: Percutaneous tracheostomy; Intensive Care Unit; Ineffective Airway Clearance; Weaning failure
MeSH Terms: conditions — Nervous System Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- critical ill patients: The investigator will enroll all the critical ill patients undergoing percutaneous tracheostomy performed in ICU
  Interventions: Procedure: Percutaneous tracheostomy

INTERVENTIONS:
Procedure: Percutaneous tracheostomy — Percutaneous tracheostomies will be performed with the kit commercially available in the current clinical practice.

SUMMARY:
Tracheostomy is worldwide performed in Intensive Care Unit (ICU). According to the current literature, indication for percutaneous tracheostomy (PDT) in ICU are: difficult prolonged weaning, prolonged mechanical ventilation, loss of airway reflex, copious secretions, upper airway obstruction. Many studies have focused on the comparison between different PDT techniques and complication. The aim of our study is to evaluate the procedural features, complications, ICU mortality, quality of life, post-discharge mortality of patients undergoing different PDT techniques performed in ICU.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* indication for tracheostomy

Exclusion Criteria:

* infectious disease of neck

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criticall ill patients requiring percutaneous tracheostomy in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-02 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety of percutaneous tracheostomy | at the beginning and at the end of the procedure

SECONDARY OUTCOMES:
Early complications | in the first 24 hours from the end of the procedure
  Early complications are:multiple intubation attempts (more than 1), accidental extubation, paratracheal insertion, injuries to blood vessels in the neck, oesophageal injury, accidental decannulation, malposition of the tracheostomy tube, tracheal cuff puncture, multiple punctures (more than 1), surgical conversion and percutaneous tracheostomy failure, minor bleeding (compressible), major bleeding (incompressible), pneumothorax
Late complications | from the 2nd day ofter the procedure until the ICU discharge (expected average of 2 weeks)
  Late complications are: minor bleeding (compressible), major bleeding (incompressible) tracheostomy puncture site infection, subglottic stenosis, fracture of a tracheal cartilage, granuloma.
Quality of life | at 3, 6 and 12 months after tracheostomy
  The investigator will use the EURO-QOL
Evaluation of organ function | At 3, 6 , and 12 months after tracheostomy
  The investigator will perform a flexible fiberoptic laryngoscopy.
Quality of voice | At 3,6, 12 months after tracheostomy
  the investigator will use a KAY elemetrics analyzer.
Mortality | at 3, 6 and 12 months from tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, Principal Investigator — Universita degli Studi di Genova
Locations (1):
- University of Genoa, Genoa, Italy, Italy